CLINICAL TRIAL: NCT01723176
Title: Evaluating Critical Care Echocardiography in Patients With Cardiopulmonary Failure at the Time of Presentation
Brief Title: Evaluation of Ultrasound of the Heart in Patients With Low Blood Pressure
Status: Withdrawn | Type: Observational
Why Stopped: study never got off the ground, no pts ever recruited
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Justin Weiner, Chief Fellow, Pulmonary and Critical Care, Northwell Health
Other Study IDs: 11-408A
Record Dates: First submitted 2012-11-01; First posted 2012-11-07 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Cardiopulmonary Failure
Keywords: goal-directed echocardiography; cardiopulmonary failure; critical care ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients in Cardiopulmonary Failure: patients in cardiopulmonary failure
  Interventions: Procedure: Echocardiography

INTERVENTIONS:
Procedure: Echocardiography

SUMMARY:
Hypothesis: Goal-directed echocardiography by trained critical care physicians is equivalent to that of echocardiography technicians/cardiologists for the purpose of determining etiology (reason) of cardiopulmonary failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present to the medical intensive care unit with cardiopulmonary failure

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to the medical intensive care unit with cardiopulmonary failure
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Assessment of left ventricular function | within four hours of ICU admission
  Will the assessment of left ventricular function by critical care physicians and echo techs be concordant?

SECONDARY OUTCOMES:
Presence of Pericardial Effusion and Severity | within 4 hrs of ICU admission
  Will the presence of pericardial effusion and severity from critical care physicians and echo techs be concordant?

OTHER OUTCOMES:
Right ventricle dysfunction | within 4 hrs of ICU admission
  Will presence of RV dysfunction with critical care physicians versus echo techs/cardiologists be concordant in our population?

CONTACTS AND LOCATIONS:
Overall Officials: Justin Weiner, DO, Principal Investigator — NS-LIJ Health System
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States